CLINICAL TRIAL: NCT05916599
Title: Evaluation of Ultrasound on Peroperative Fluid Management in Patients Undergoing Hip Surgery Under Spinal Anesthesia
Brief Title: Ultrasound in Evaluation of Preoperative Fluid Management of Hip Fracture Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Döndü Genc Moralar, head of anesthesiology, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 138
Record Dates: First submitted 2023-05-03; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Lung Edema; Hip Fractures
MeSH Terms: conditions — Pulmonary Edema; Hip Fractures | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Goal directed: The inferior vena cava collapse index IVC CI and lung ultrasound score (LUS) measurements and goal directed fluid therapy will be done.Patients in the group will be started with fluid replasment at an hourly rate of 2ml/kg/h and with ultrasound measurement the infused fluid will be evaluated and regulated.
  Interventions: Device: ultrasound
- conventional: . Group applying zero balance liquid therapy to patients with conventional methods is planned. Crystalloid liquid infusion at a rate of 2ml/kg/hour will be administered to the patients in the group additional fluid replacement will be decided by monitoring bleeding and urinary output, zero balance is aimed at patients.

INTERVENTIONS:
Device: ultrasound — a device which is used in intensive care units,
  Groups: Goal directed

SUMMARY:
Goal directed fluid therapy is a new standard surgical procedure which is successful in patients undergoing hip revision arthroplasty, There has been a reduction of postoperative complications, most importantly surgery with a decrease inbleeding, as well as in hospital and intensive care stays it is related. The aim of this study is to evaluate effectiveness of pulmonary ultrasound score and vena cava collapse index measurements in the patients undergoing hip surgery under spinal anesthesia and relation with peroperative fluid management.

DETAILED DESCRIPTION:
Patients who will undergo hip surgery under spinal anesthesia using the closed envelope method it will be randomized and divided into 2 groups.

1.The inferior vena cava collapse index IVC CI and lung ultrasound score (LUS) measurements and goal directed fluid therapy will be done 2. Group applying zero balance liquid therapy to patients with conventional methods is planned.

1. Patients in the group will be started with fluid replasment at an hourly rate of 2ml/kg/h and with ultrasound measurement the infused fluid will be evaluated and regulated.
2. Crystalloid liquid infusion at a rate of 2ml/kg/hour will be administered to the patients in the group additional fluid replacement will be decided by monitoring bleeding and urinary output, zero balance is aimed at patients. Both groups were treated with spinal anesthesia in the postoperative period 120. minute IVC CI and the LUS score value will be checked.

If the CI is below 50% and the LUS score is below 15, fluid management will be considered as successful.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 65 who will undergo hip surgery
* ASA I-II-III patients

Exclusion Criteria:

* Patients under the age of 65
* Patients with ASA IV-V
* Patients with BMI>above 35
* Patients with an Lus score of 15 and above
* Patients who have not undergone spinal anesthesia

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients undergoing hip surgery under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-08-09 (Estimated); Study Completion 2023-09-12 (Estimated)

PRIMARY OUTCOMES:
comparison of groups for change of vena cava inferior collapsibility index in 4 time frames | vena cava inferior collapsibility index measurements will be done in 4 time frames.1.just before spinal anesthesia, 2. at fifth minute of surgery ,3. at 15. minute of surgery, 4 immediatelyafter surgery
  vena cava inferior collapsibility index will be measured at 4 time frames by using ultrasound,changes over 20% will be considered as significant

SECONDARY OUTCOMES:
comparison of groups for pulmonary edema | measurements will be done in 4 time frames.1.just before spinal anesthesia, 2. at fifth minute of surgery ,3. at 15. minute of surgery, 4immediately after surgery
  detecting 12 parts of lung with ultrasound with a score of 1-36

CONTACTS AND LOCATIONS:
Overall Officials: zuhal çavuş, MD, Principal Investigator — gaziosmanpasa TREH
Locations (1):
- Gaziosmanpasa Education and Research Hospital, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)